CLINICAL TRIAL: NCT01650987
Title: Prospective Observational Study of Toxicities of Cervix and Corpus Uteri Carcinomas Treatment and Evaluation of Impact on Sexual Function
Brief Title: Toxicities of Cervix and Corpus Uteri Carcinomas Treatment and Evaluation of Impact on Sexual Function
Acronym: SEXUTOX
Status: Completed | Type: Observational
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Other Study IDs: SEXUTOX
Record Dates: First submitted 2012-07-20; First posted 2012-07-26 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Corpus Uteri Carcinoma
Keywords: carcinoma; uterus; Not metastatic
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Col 1: Patient with uterus adenocarcinoma, treated by surgery, then surveillance without complementary treatment
- Col 2: Patient with uterus adenocarcinoma, treated by surgery then adjuvant radiotherapy
- Col 3: patient with uterus adenocarcinoma, treated by surgery then curietherapy of vaginal dome
- Endometrial 4: patient with cervix carcinoma stage IA2 to IIB, treated by surgery only
- endometrial 5: patient with cervix carcinoma stage IA2 to IIB, treated by surgery then curietherapy
- endometrial 6: patient with cervix carcinoma stage IA2 to IIB, treated by surgery then curietherapy and radiotherapy

SUMMARY:
Evaluate the toxicities of cervix and corpus uteri carcinomas treatment

DETAILED DESCRIPTION:
Evaluate the toxicities of cervix and corpus uteri carcinomas treatment on sexual function after treatment (radiotherapy and/or surgery)

ELIGIBILITY:
* Inclusion Criteria:
* Patients whose treatment is provided to Centre Oscar Lambret
* With a corpus uteri adenocarcinoma, no metastatic, treated by:
* Surgery and observation without complementary treatment
* Or surgery and adjuvant radiotherapy
* Or Surgery and curietherapy of vaginal dome
* With a cervix carcinoma, stade IA2 to IIB proximal, treated by :
* External radiochemotherapy and curietherapy
* Or only surgery
* Or pre-surgical curietherapy and surgery
* Age > 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with a corpus uteri carcinoma, without metastasis.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2009-05; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Toxicities including on sexual function | up to 3 years
  According to Lent-Soma, NCICTC-AE v3.0, Franco-Italian Glossary

SECONDARY OUTCOMES:
Compare the various scales of toxicity | up to 3 years
  Compare the various scales of toxicity
Study the sexual behavior modifications | up to 3 years
  According to a questionnaire and a personal discussion
Specify correlation modifications of sexual behavior | up to 3 years
  Specify the existence of a correlation between toxicities included modifications and sexual behavior modifications

CONTACTS AND LOCATIONS:
Overall Officials: Philippe NICKERS, MD, Study Director — Oscar Lambret Center
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: No